CLINICAL TRIAL: NCT05792644
Title: The Therapeutic Effect of Crizotinib in Patients With ALK-rearrangement-negative But High Expression of ALK Phosphorylation
Brief Title: Therapeutic Effect of Crizotinib for Rearrangement-negative, High Phosphorylated ALK Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Xuemeng Li, Clinical Doctor, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XLi
Record Dates: First submitted 2022-09-18; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: ALK Phosphorylation
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Intervention Model Description: Some patients with histologically or cytologically confirmed stage IIIB or IV ALK-negative non-small-cell lung cancer (NSCLC) participated in this study following the failure of initial treatments. The ALK phosphorylation expression was detected in histologic samples of patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patients with positive ALK phosphorylation expression were treated with crizotinib 250 mg/day orally. A treatment cycle was defined as 30 days of once-daily crizotinib treatment. Treatment with crizotinib continued until the patient experienced unacceptable toxicity, was pregnant, or started new cancer therapy.
  Interventions: Drug: crizotinib for rearrangement-negative, high phosphorylated ALK patients

INTERVENTIONS:
Drug: crizotinib for rearrangement-negative, high phosphorylated ALK patients — Patients with positive ALK phosphorylation expression were treated with crizotinib 250 mg/day orally. A treatment cycle was defined as 30 days of once-daily crizotinib treatment. Treatment with crizotinib continued until the patient experienced unacceptable toxicity, was pregnant, or started new cancer therapy.

SUMMARY:
Patients with histologically or cytologically confirmed stage IIIB or IV ALK-negative non-small-cell lung cancer (NSCLC) participated in this study following the failure of initial treatments. The ALK phosphorylation expression was detected in histologic samples of patients. patients with positive ALK phosphorylation expression were treated with crizotinib .

DETAILED DESCRIPTION:
Some patients with histologically or cytologically confirmed stage IIIB or IV ALK-negative non-small-cell lung cancer (NSCLC) participated in this study following the failure of initial treatments. The ALK phosphorylation expression was detected in histologic samples of patients. patients with positive ALK phosphorylation expression were treated with crizotinib 250 mg/day orally. A treatment cycle was defined as 30 days of once-daily crizotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 80 years
2. Histologically or cytologically confirmed stage IIIB or IV ALK-negative NSCLC by NGS
3. Disease staging determined according to the International Association for the Study of Lung Cancer 8th edition TNM staging system
4. All measurable Response Evaluation Criteria in Solid Tumors (RECIST) target lesions
5. Treatment failure at the end of the most recent treatment episode
6. World Health Organization/Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Consent of patients for participation in this study
8. Complete clinical data
9. High ALK phosphorylation level

Exclusion Criteria:

1. Patients with cognitive impairment, severe psychiatric diseases, or other disorders likely to impact informed consent
2. Patients with uncontrolled systemic disease
3. Patients with other malignant tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy | SIx months
  The clinical efficacy was evaluated according to the RECIST 1.1 guidelines[5], including PD, stable disease (SD), partial response (PR), and complete remission (CR), where the objective response rate (ORR) = (CR + PR) number of cases/total number of cases, and the disease control rate (DCR) = (CR + PR + SD) number/total number of cases.

SECONDARY OUTCOMES:
The progression-free survival | 3 years
  The progression-free survival (PFS) was defined as the time from the date of first treatment to any recurrence or last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China